CLINICAL TRIAL: NCT00138437
Title: Molecular Epidemiology of Leprosy in Colombia
Brief Title: Molecular and Immunological Tools for Detection of Strain Diversity, Drug Resistance and Immunological Responses
Status: Completed | Type: Observational
Sponsor: Colorado State University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09-817H
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Leprosy
Keywords: leprosy; Colombia
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, Nasal Swabs, Skin Biopsies and scrapings
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Leprosy Patients (Group 1): All leprosy patients
- Household Contacts (Group 2): Household contacts with known contact with leprosy patients
- Healthy Individuals (Group 3): Healthy persons with no known contact with leprosy patients

SUMMARY:
The purpose of this study is to determine what factors contribute to the continued incidence of leprosy in Colombia. Study participants will include volunteering and consenting individuals, older than 4 years of age, representing three study groups:

1. healthy persons with no known contact with leprosy patients
2. patients reporting at Instituto Colombiano de Medicina Tropical-CES and Impresa Social del Estado Sanatorio Agua de Dios with a new diagnosis of leprosy or relapse of leprosy
3. household contacts of leprosy patients described in group 2. Blood, nasal swabs, slit skin smears, and biopsies will be taken from the volunteers to learn the strains of leprosy-causing bacteria in the area, the immune responses (body's response to disease) in local residents against the bacteria, and the pattern of leprosy transmission. Individuals will participate in this study for 1-10 days, and the study will last for 3 years.

DETAILED DESCRIPTION:
The overall objectives of this study are to understand the factors leading to continued incidence of leprosy in Colombia by novel molecular methodologies using a combination of retrospective and prospective sampling approaches using three study groups. Specific objectives are: (1) strain typing of M. leprae isolates obtained from newly diagnosed leprosy patients and household contacts (HHCs) in Colombia to identify clusters and transmission patterns when combined with conventional epidemiological criteria; (2) to determine the viability of M. leprae by mRNA detection in specimens collected from new leprosy patients and HHCs; (3) to identify and determine the extent of mutations conferring resistance in past and circulating M. leprae isolates from leprosy patients to two Multidrug therapy (MDT) drugs; dapsone and rifampicin; (4) to detect chains of transmission in endemic populations by a retrospective analyses of isolates in sample banks when combined with strain typing information from new cases and conventional epidemiological criteria; and (5) to detect, compare, and delineate immune response profiles to M. leprae antigens as biomarkers for early detection of leprosy and prediction of clinical outcome (susceptible, infected, and resistant individuals) among three study groups. Study participants for prospective sample collections will include volunteering and consenting individuals older than 4 years of age, representing three study groups: (1) healthy persons with no known contacts with leprosy patients, (2) patients reporting at Instituto Colombiano de Medicina Tropical-CES (ICMT-CES) and Impresa Social del Estado Sanatorio Agua de Dios for the diagnosis of leprosy and/or relapse of leprosy, and (3) household contacts (HHC) of leprosy patients reporting at Instituto Colombiano de Medicina Tropical-CES (ICMT-CES) and Impresa Social del Estado Sanatorio Agua de Dios. Blood, nasal swabs, slit skin smears and biopsies will be obtained prospectively from individuals greater than 4 years of age representing three study groups: newly diagnosed and relapse leprosy patients, their household contacts; and healthy persons with no known contacts with leprosy patients. Retrospective archived samples from past and present leprosy patients will be included when available. DNA and RNA based methodologies will be developed and applied to obtain data necessary for substantiation of a number of factors implicated in transmission of leprosy in Colombia. Nucleic acid based molecular methods like Multiple Locus Variable number of tandem repeat Analysis (MLVA) and Single Nucleotide Polymorphisms (SNPs) will be performed for strain typing M. leprae, in combination with epidemiological information to delineate the distribution of types of the organism in various regions of Colombia. Other DNA markers such as mutations causing drug resistance will also be collected from the M. leprae containing specimens. Due to the lack of methods to cultivate M. leprae, viability of the organism in newly collected biological samples will be tested by mRNA detection. A database will be generated which will include M. leprae genotypes, patient history (clinical and demographic) for comprehensive epidemiological analyses to monitor prevailing M. leprae population structures reflective of short and long range dissemination; and correlations between disease type and genotype; to track evolutionary and transmission patterns. Profiling of host immunological responses during infection with M. leprae will be done by detection of a panel of cytokines at the level of mRNA and/or protein, and detection of antibodies against M. leprae antigens in leprosy patients, their household contacts and healthy individuals with no known history or contacts with leprosy patients.

ELIGIBILITY:
Inclusion Criteria:

* All leprosy patients (Group1), their household contacts (Group 2) and healthy persons with no known contacts with leprosy patients (Group 3), between the ages of 18 and 70 years willing to participate in this study.

Exclusion Criteria:

* Patients unwilling to participate or unable to give informed consent will be excluded from the study.
* Pregnant women will be excluded.

Exclusion criteria for objective A.5 are one or more of the following conditions:

* Chronic illnesses such as cancer
* Diabetes
* Hepatitis
* HIV
* Tuberculosis
* Undergoing corticosteroid therapy
* Current or previous history of immunosuppressive therapy as assessed from medical records and interviews with a physician.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants for prospective sample collections will include volunteering and consenting individuals older than 18 years of age, representing three study groups
Sampling Method: Non-Probability Sample
Enrollment: 1554 (Actual)
Dates: Start 2006-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Strain typing: identification of genotypes | Dec, 2010

CONTACTS AND LOCATIONS:
Overall Officials: Varalakshmi Vissa, PhD, Principal Investigator — Colorado State University; Nora Cardona-Castro, MD, MSc, Principal Investigator — Instituto Colombiano de Medicina Tropical - Universidad CES
Locations (2):
- Colombia (2):
  - Impresa Socail del Estado Sanatorio Agua de Dios, Agua de Dios
  - Instituto Colombiano de Medicina Tropical-CES, Sabaneta